CLINICAL TRIAL: NCT00589615
Title: Effectiveness of an Educational Program in the Prevention of Osteoporosis and Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Miina Sillanpää Foundation (Unknown)
Responsible Party: Matti Välimäki, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 325/E05/01; Miina Sillanpää Foundation
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2008-01-10 (Estimated); Status verified 2007-12

CONDITIONS: Fractures; Osteoporosis
Keywords: vitamin D; bone density
MeSH Terms: conditions — Fractures, Bone; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The multidisciplinary osteoporosis prevention study started with a five-day program at a rehabilitation centre and will be followed by one-day group appointments twice.
  Interventions: Behavioral: multidisciplinary osteoporosis prevention educational program
- 2 (No Intervention): The control group will get information about osteoporosis through media and health care system.

INTERVENTIONS:
Behavioral: multidisciplinary osteoporosis prevention educational program — The program includes individualized counseling aimed at improving diet, muscle strength, balance, and informing individuals about home hazards and the use of medicine.
  Arms: 1

SUMMARY:
The study will elucidate the effectiveness of an educational program in the prevention of osteoporosis and fractures. A random sample of the female population in Southern Finland (Uusimaa region) within the age group of 60-70 years was drawn from the population registry. From 1996 through 2000, 2181 women from the population register were recruited and randomly assigned to the intervention and to the control group. The subjects in the intervention group have been on a multidisciplinary program and the subjects in the control group received osteoporosis prevention information through the media and health care system. An end point is any fracture during the ten-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-70 years and living in southern Finland (Uusimaa region)

Ages: 60 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2181 (Actual)
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: Matti J Välimäki, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Miina Sillanpää Foundation, Helsinki, Finland

REFERENCES:
- [Background] Evio S, Pekkarinen T, Sintonen H, Tiitinen A, Valimaki MJ. The effect of hormone therapy on the health-related quality of life in elderly women. Maturitas. 2007 Feb 20;56(2):122-8. doi: 10.1016/j.maturitas.2006.06.009. Epub 2006 Dec 8. PMID 17158003
- [Background] Enattah N, Pekkarinen T, Valimaki MJ, Loyttyniemi E, Jarvela I. Genetically defined adult-type hypolactasia and self-reported lactose intolerance as risk factors of osteoporosis in Finnish postmenopausal women. Eur J Clin Nutr. 2005 Oct;59(10):1105-11. doi: 10.1038/sj.ejcn.1602219. PMID 16015262